CLINICAL TRIAL: NCT01546636
Title: The Effect of Ventilation on Cerebral Oxygenation in the Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Cardiac Anesthesia and Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EH10-184
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Results first posted 2013-12-17 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Cerebral Ischemia
Keywords: Cerebral desaturation events; Cerebral oximetry; Beach chair position
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypocapnic group (Placebo Comparator): Patients will be ventilated to an ETCO2 of 30-32 mm Hg.
  Interventions: Other: Hypocapnic group
- Normocapnic group (Active Comparator): Patients will be ventilated to an ETCO2 of 40-42 mm Hg
  Interventions: Other: Normocapnic group

INTERVENTIONS:
Other: Hypocapnic group — Patients will be ventilated to an ETCO2 of 30-32 mm Hg.
  Arms: Hypocapnic group
Other: Normocapnic group — Patients will be ventilated to an ETCO2 of 40-42 mm Hg
  Arms: Normocapnic group

SUMMARY:
The aim of this clinical investigation is to determine the effect of intraoperative ventilation on cerebral oxygen saturation in patients undergoing arthroscopic shoulder surgery in the beach chair position (BCP)

DETAILED DESCRIPTION:
Recent developments in near-infrared spectroscopy technology now permit rapid assessment of cerebral oxygenation (SctO2) using non-invasive probes. A high incidence cerebral desaturation events (CDE-defined as a decrease in SctO2 values below 20% of baseline measures or absolute SctO2 values ≤ 55 for ≥ 15 seconds) have been observed in previous investigation of patients undergoing shoulder surgery in BCP with hyperventilation. The investigators hypothesize that the incidence of CDE will be reduced in patients ventilated at normocapnic levels (end-tidal carbon dioxide values (ETCO2) of 40-42 mm Hg) when compared to subjects hyperventilated (ETCO2 of 30-32 mm Hg) in the operating room. Patients undergoing shoulder surgery in the BCP will be randomized to a hypocapnic group (ETCO2 of 30-32 mm Hg) or a normocapnic group (ETCO2 of 40-42 mm Hg). Cerebral oxygenation will be measured continuously throughout the procedure to assess perioperative SctO2 values and the incidence of CDE. The investigators previously observed an association between CDE in the operating room and postoperative nausea and vomiting. Therefore, the effect of ventilatory pattern and intraoperative SctO2 on clinical recovery will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective shoulder arthroscopy under general anesthesia in the BCP.

Exclusion Criteria:

* Exclusion criteria include 1) history of pre-existing cerebrovascular disease or orthostatic hypotension 2) age < 18 years 3) American Society of Anesthesiologists Physical Status IV or V.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

REFERENCES:
- [Derived] Murphy GS, Szokol JW, Avram MJ, Greenberg SB, Shear TD, Vender JS, Levin SD, Koh JL, Parikh KN, Patel SS. Effect of ventilation on cerebral oxygenation in patients undergoing surgery in the beach chair position: a randomized controlled trial. Br J Anaesth. 2014 Oct;113(4):618-27. doi: 10.1093/bja/aeu109. Epub 2014 May 23. PMID 24860157

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 70 patients presenting for elective shoulder surgery at NorthShore University HealthSystem were enrolled in the clinical trial.
Pre-assignment Details: All enrolled participants completed the study, and complete data was collected on all subjects.
Period: Overall Study
Arm/Group | Hypocapnic Group | Normocapnic Group
Started | 36 | 34
Completed | 36 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants was determined by performing a sample size calculation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypocapnic Group | Normocapnic Group | Total
Number analyzed (Participants) | 36 | 34 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 30 | 61
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (13.8) | 54.7 (12.4) | 53.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 50
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 36 | 34 | 70

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Cerebral Desaturation Events
Description: Cerebral desaturation events were measured with near-infrared spectroscopy
Time Frame: Intraoperative-first 2 hours
Measure: Number; unit: number of events
Arm/Group | Hypocapnic Group | Normocapnic Group
Number analyzed (Participants) | 36 | 34
number of events | 19 | 3

2. Secondary Outcome: Number of Patients Experiencing Nausea and Vomiting
Description: Assessed by recovery nurses
Time Frame: Postanesthesia care unit-first 2 hours
Measure: Number; unit: participants
Arm/Group | Hypocapnic Group | Normocapnic Group
Number analyzed (Participants) | 36 | 34
participants | 12 | 3

3. Secondary Outcome: Postanesthesia Care Unit Length of Stay (Total Time)
Time Frame: Approximately 5 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | Hypocapnic Group | Normocapnic Group
Number analyzed (Participants) | 36 | 34
minutes | 81.5 [23 to 267] | 69 [19 to 133]

ADVERSE EVENTS:
Time Frame: Until the time of hospital discharge
Description: Patients were followed until hospital discharge
Arm/Group | Hypocapnic Group | Normocapnic Group
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34
Other Adverse Events (participants affected / at risk) | 0/36 | 0/34

LIMITATIONS AND CAVEATS:
There were no technical limitations to the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes